CLINICAL TRIAL: NCT02978664
Title: The Impact of Distraction on Adenoma Detection Rate in Patients Undergoing Colonoscopy With Air Insufflation, Water Immersion and Water Exchange
Brief Title: The Impact of Distraction on Adenoma Detection Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DalinHsieh201401
Record Dates: First submitted 2016-04-08; First posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Adenoma
Keywords: colonoscopy; water exchange; adenoma detection rate; distraction
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Air insufflation (Active Comparator): Air insufflation will be used throughout whole procedure of colonoscopy
  Interventions: Procedure: Air insufflation
- water immersion (Active Comparator): Water will be infused during the insertion phase and removed during withdrawal phase of colonoscopy
  Interventions: Procedure: water immersion
- water exchange (Active Comparator): Water will be infused and removed during insertion phase of colonoscopy
  Interventions: Procedure: Water exchange

INTERVENTIONS:
Procedure: Air insufflation — Air insufflation during colonoscopy including insertion phase
  Arms: Air insufflation
Procedure: water immersion — Water will infused during insertion phase and removed during withdrawal phase of colonoscopy.
  Arms: water immersion
Procedure: Water exchange — Water will infused and removed during insertion phase of colonoscopy
  Arms: water exchange

SUMMARY:
The investigators will review video-recordings of three randomized, controlled trials (NCT01535326, 01699399, and 01894191) comparing air insufflation, water immersion and water exchange during colonoscopy. These studies were all conducted at Buddhist Dalin Tzu Chi Hospital.

DETAILED DESCRIPTION:
The investigators will review video-recordings of three randomized controlled trials (NCT01535326, 01699399, and 01894191) comparing air insufflation, water immersion and water exchange. These studies were conducted at Buddhist Dalin Tzu Chi Hospital. Permission will be obtained from the local Institutional Review Board (IRB) to review, analyze and report de-identified findings.

Two experienced endoscopists (YHH and CWT) performed all the recorded colonoscopies. Recordings will be selected for review if they are complete examinations; include clear identification of the appendiceal orifice and/or the ileocecal valve, indicating arrival at the cecum; available in the appropriate format for video editing; and contain no patient or endoscopist identifiers. Patients with incomplete recordings and a history of bowel resection will be excluded from analysis. The included video recordings will be edited to remove the insertion phase to blind the study reviewer to the insertion techniques. One blinded reviewer uninvolved in the performance of the colonoscopies will be in charge of evaluating the selected videos, using the criteria described by Yung et al

ELIGIBILITY:
Inclusion Criteria:

* if they are complete examinations; include clear identification of the appendiceal orifice and/or the ileocecal valve, indicating arrival at the cecum; available in the appropriate format for video editing; and contain no patient or endoscopist identifiers.

Exclusion Criteria:

* Patients with incomplete recordings and a history of bowel resection will be excluded from analysis.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate | one week after colonoscopy

SECONDARY OUTCOMES:
Distraction score | Immediate after video reviewing
Withdrawal technique as specified by Lee RH (citation 1) | immediate after video reviewing
  adequacy of distention (0-5), fold examination (0-5) and cleaning (0-5) for each colonic segment
Bowel preparation score | immediate after video reviewing
  Boston bowel preparation score

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsi Hsieh, MD, Principal Investigator — Dalin Tzu Chi General Hospital
Locations (1):
- Buddhist Dalin Tzu Chi General Hospital, Chiayi City, Taiwan, Taiwan

REFERENCES:
- [Background] Lee RH, Tang RS, Muthusamy VR, Ho SB, Shah NK, Wetzel L, Bain AS, Mackintosh EE, Paek AM, Crissien AM, Saraf LJ, Kalmaz DM, Savides TJ. Quality of colonoscopy withdrawal technique and variability in adenoma detection rates (with videos). Gastrointest Endosc. 2011 Jul;74(1):128-34. doi: 10.1016/j.gie.2011.03.003. Epub 2011 Apr 30. PMID 21531410
- [Background] Leung FW. Water exchange may be superior to water immersion for colonoscopy. Clin Gastroenterol Hepatol. 2011 Dec;9(12):1012-4. doi: 10.1016/j.cgh.2011.09.007. Epub 2011 Sep 22. No abstract available. PMID 21946120
- [Background] Yung VY, Yen AW, Leung JW, Mann SK, Wilson MD, Leung FW. Validation of a novel method for analyzing video recordings of the withdrawal phase of air insufflation and water exchange colonoscopy - documentation of distractions from focused mucosal inspection. J Interv Gastroenterol. 2014 Jan;4(1):8-12.
- [Derived] Hsieh YH, Koo M, Tseng CW, Yang HW, Leung FW. Reduction of multitasking distractions underlies the higher adenoma detection rate of water exchange compared to air insufflation - blinded analysis of withdrawal phase videos. United European Gastroenterol J. 2019 Mar;7(2):230-238. doi: 10.1177/2050640618817105. Epub 2018 Dec 5. PMID 31080608